CLINICAL TRIAL: NCT04329013
Title: The Comparison of Left Lateral Versus Prone Position in Saliva Droplet Spreading During Upper Gastrointestinal Endoscopy; a Pilot Study of Randomized Trial
Brief Title: Position of EGD in Droplet Spreading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RP017
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Cotamination on Face Shield

STUDY DESIGN:
Intervention Model Description: We will randomize the patients who need EGD into 2 groups; left lateral and prone position by block of 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left lateral position (Active Comparator): The patient will be in left lateral position during EGD
  Interventions: Other: Left lateral Position during intervention
- Prone position (Experimental): The patient will be in prone position during EGD
  Interventions: Other: Prone Position during intervention

INTERVENTIONS:
Other: Left lateral Position during intervention — Left lateral position during EGD
  Arms: Left lateral position
Other: Prone Position during intervention — Prone position during EGD
  Arms: Prone position

SUMMARY:
The association between position of upper gastrointestinal endoscopy (EGD) and saliva droplet spreading has never been studied. In the era of contagious viral spreading, this pilot study is aimed to assess adenosine triphosphate (ATP) at the face shield of endoscopist which can represent the saliva droplet spreading of patients in left lateral and prone position during EGD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have the indication for upper gastrointestinal endoscopy

Exclusion Criteria:

* Cannot be in prone position
* The endoscopist deny the assigned position in any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The level of adenosine triphosphate (ATP) on face shield of endoscopist | immediately following the procedure
  Measuring the ATP on face shield of endoscopist by using ATP luminometer. It is measured in relative light unit (RLU). The level of ATP is concordant with the level of bacteria on that measuring object.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Do not plan for data sharing due to the privacy of each patient.